CLINICAL TRIAL: NCT05273203
Title: A Proposed Design for a Dose-Response Clinical Trial in High Risk Adults
Brief Title: The Influence of Football Training as a medicine_FIM_UTH
Acronym: FIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Ioannis G. Fatouros, Professor, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FIM_UTH
Record Dates: First submitted 2022-02-16; First posted 2022-03-10 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Soccer Training; Body Composition; Physical Activity; Healthy
Keywords: Football; Health; Performance; Somatometric; Quality of life
MeSH Terms: conditions — Motor Activity | interventions — fim 1; fim 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Experimental): No intervention. Participated only in measurements at baseline and at 6 months.
  Interventions: Behavioral: Control
- FIM-1 (Experimental): Participated in a supervised 6 months football training program once per week and in measurements at baseline and at 6 months.
  Interventions: Behavioral: FIM-1
- FIM-2 (Experimental): Participated in a supervised 6 months football training program twice per week and in measurements at baseline and at 6 months.
  Interventions: Behavioral: FIM-2
- FIM-3 (Experimental): Participated in a supervised 6 months football training program thrice per week and in measurements at baseline and at 6 months.
  Interventions: Behavioral: FIM-3

INTERVENTIONS:
Behavioral: FIM-1 — A football group (12 participants/session) will participate in 60 minutes football training that will contain warm-up, football technical drills and exercises, fitness exercises and football game.
  Other Names: Football training
  Arms: FIM-1
Behavioral: FIM-2 — A football group (12 participants/session) will participate in 60 minutes football training that will contain warm-up, football technical drills and exercises, fitness exercises and football game.
  Other Names: Football training
  Arms: FIM-2
Behavioral: FIM-3 — A football group (12 participants/session) will participate in 60 minutes football training that will contain warm-up, football technical drills and exercises, fitness exercises and football game.
  Other Names: Football training
  Arms: FIM-3
Behavioral: Control — No football training will be performed during 6 months period. Participation only in measurements at baseline and at 6 months.
  Arms: Control

SUMMARY:
The purpose of this randomized controlled study will be to inestigate the relationship between recreational football training at various training volumes and the health responses of middle-aged participants at high risk for metabolic and / or cardiovascular disease.

DETAILED DESCRIPTION:
A controlled, randomized, four-group, repeated-measures clinical trial will be apllied. Males and females middle-aged volunteers (age 40-60 years) will participate in the present study. The participants will not suffer from any musculoskeletal injuries that will limit their ability to perform the exercise protocols.

The study will be consisted of the following stages:

1. In the first phase all participants will sign an informed consent form after they will be informed about all benefits and risks of this study and they will sign a recent historical of musculoskeletal injury or illness form.
2. Initial testing: body weight (BW) and height, BMI, electrocardiogram (ECG), RMR, daily physical activity (PA) and daily nutritional intake (participants will be instructed by a dietitian how to record a 7 days diet recalls).
3. A 4-week adaptive period: based on a dietary analysis, participants will be given a dietary plan (considering the RMR and total daily physical activity related energy expenditure), providing an isocaloric diet over the initial 4-week adaptive period and during study. During this adaptive period, volunteers will also be familiarized with exercises techniques and overload patterns that will be used throughout the study through 4 preparatory sessions.
4. At the end of the adaptation period, participants will participate in assessment procedures (baseline testing) at University facilities. Fasting blood samples will be collected by venipuncture using a disposable needle (20-gauge) in order to etsimate the lipid profile (TCHO, LDL, HDH, TG), fasting glucose and insulin, Hemoglobin (HbA1c) test in order to measure the amount of blood sugar (glucose) attached to hemoglobin and HOMA-IR, muscle damage markers (CK), inflammation markers (WBC and GRA), oxidative stress markers (PC, GSH, GSSG, ΤΑC and CAT), cortisol, blood test (HGB, HCT, LYM, MON, PLT and RBC) and cytokines indicators (IL-1b, IL-6 and CRP). The following will be included in the assessment procedures: Body weight (BW) and Height, body mass index (BMI), Body composition (DXA method), the circumferences of waist and hip in order to estimate the waist hip ratio (WHR). Also, the volunteers will participate in health-related measurements as: Bone mineral density, Bone mineral content, Hip structural analysis, Arterial blood pressure- Mean arterial blood pressure, resting heart rate, ultrasonography for heart and blood vessels and functional movement screen (FMS). The performance measurements in baseline testing are included the following procedures: maximal oxygen consumption and heart rate maximum (Vo2max-HRmax prediction using the Balke test), strength (1- repetition maximum in leg press and chest press), the knee-hip and ankle range of motion will be determined using a goniometer, the balance and gait speed indicator will be determine using Romberg's test and short physical performance battery tool respectively. Also, muscle endurance tests will be used and flexibility will be measured using sit and reach test. 10m and 30m sprint test will be measured in the same period using photocells device and the conter movement jump will be measured using a force platform. Measurements of well-being (vitality, quality of life, flow, depression, behavioral regulations in exercise and pgycological well being) will be performed using modified questionnaires.
5. After the adaptive period all participants will be randomly assigned to four groups (control, 1 session/week, 2 sessions/week, 3 sessions/week). The footbal training that will be used throughout the 6 months intervention will be consisted of wurm up (7-10 minutes), Tecnhical drills (5-8 minutes), fitness exercises (5-10 minutes), football games (30 minutes) and recovery period (5 minutes). During the sessions will be assessed the change in Heart rate using a heart rate monitor and the field activity will be recorded using a global positiong system (GPS). At the end of every session will be used Borg scale in monitoring progress and mode of exercise. Also, following a single training session both at pre and post training will be measured the delayed onset muscle soreness scale (DOMS), the Creatine Kinase activity, the isometric force of knee extensors and knee flexors, the eccentric and concentric peak torque using isokinetic dynamometer, the counter movement jumb ability and blood samples will be collected in order to estimate biochemical indicators (Oxidative stress and inflammatory response). Fianlly, the energy expenditure during training will be measured via blood lactate and oxygen consumption.
6. After 6 months of football intervention all participants will participate in assessment procedures (post-training testing) at University facilities within 5 days after the completion of the last training session.

All participants will be randomly assigned to the following four groups:

1. Control group (no training)
2. FIM-1 (1 session/week)
3. FIM-2 (2 sessions/week)
4. FIM-3 (3 sessions/week)

ELIGIBILITY:
Inclusion Criteria:

1. The participants Vo2max <30ml/kg/min
2. age of 40-60 years
3. medical clearance for strenuous physical training
4. Free of chronic diseases
5. Free of musculoskeletal injury
6. waist circumference 80≥ cm for female and 94≥ cm for Male participants
7. no weight loss greater >10% of body mass before (≤6 months) the study
8. no diet intervention or usage of nutritional supplements/medications before (≥6 months) and during the study

Additionaly the participants will have at least two of the following risk factors

* overweight/obese (BMI 25.0-35.0)
* Fasting Glucose≥100 mg/dl
* Blood Pressure≥120/80 mmHg
* Total Cholesterol≥190 mg/dl
* High Desnity lipoprotein< 35 mg/dl for male and < 39 mg/dl for female participants
* Low Density Lipoprotein≥100 mg/dl
* Triglycerides≥150 mg/dl

Exclusion Criteria:

Participants will be excluded from the study if they:

1. will not participate in ≥80% of total exercise sessions
2. will adhere to a nutritional intervention during the study
3. will modify the habitual physical activity levels during the study
4. Musculoskeletal injury
5. Chronic disease

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in body mass | At baseline and at 6 months
  Body mass (kg) wil be measured using a beam balance
Change in Body mass index | At baseline and at 6 months
  Body mass index wil be calculated using the Quetelet's equation
Change in Waist circumference | At baseline and at 6 months
  Waist circumference (cm) will be measured using a Gullick II tape
Change in Hip circumference | At baseline and at 6 months
  Hip circumference (cm) will be measured using a Gullick II tape
Change in Waist-to-hip ratio | At baseline and at 6 months
  Waist-to-hip ratio will be calculated by dividing the waist by the hip measurement
Change in Body fat | At baseline and at 6 months
  Body fat (%) will be assessed by whole-body dual-energy X-ray absorptiometry (DXA)
Change in fat mass | At baseline and at 6 months
  Body fat (kg) will be assessed by whole-body dual-energy X-ray absorptiometry (DXA)
Change in fat-free mass | At baseline and at 6 months
  Fat-free mass (kg) will be assessed by whole-body dual-energy X-ray absorptiometry (DXA)
Change in resting metabolic rate (RMR) | At baseline, at 6 months and 24 hours, 48 hours and 72 hours after
  RMR (kcal) will be measured using a portable open-circuit indirect calorimeter with a ventilated hood system
Change in maximal strength (1RM) | At baseline and at 6 months
  1RM (kg) for the lower body will be measured bilaterally on a horizontal leg press, while 1RM (kg) for the upper body will be measured on a horizontal chest press
Change in maximal oxygen consumption (VO2max) | At baseline and at 6 months
  VO2max (ml/kg/min) will be estimated using a low-risk submaximal treadmill walking test
Change in dietary intake | At baseline and at 6 months
  Dietary intake (kcal) will be assessed using 7-day recalls
Change in daily physical activity | At baseline and at 6 months
  Daily physical activity will be assessed accelerometry device
Change in body mass content (BMC) | At baseline and at 6 months
  BMC (g) will be assessed by dual energy X-ray absorptiometry (DXA) of the total body, hip of non-dominant and dominant limb, spine and wrist
Change in body mass density (BMD) | At baseline and at 6 months
  BMD (g) will be assessed by dual energy X-ray absorptiometry (DXA) of the total body, hip of non-dominant and dominant limb, spine and wrist
Change in hip structural analysis | At baseline and at 6 months
  hip structural analysis will be assessed by dual energy X-ray absorptiometry (DXA) of the total body, hip of non-dominant and dominant limb, spine and wrist
Change in resting systolic (SBP) and diastolic (DBP) blood pressures | At baseline and at 6 months
  Resting SBP (mmHg) and DBP (mmHg) will be assessed by a manual sphygmomanometer
Change in mean arterial pressure (MAP) | At baseline and at 6 months
  MAP (mmHg) will be calculated using the following equation : MAP = SBP + (DBP × DBP) / 3
Change in resting heart rate (RHR) | At baseline and at 6 months
  RHR will be measured by pulse palpation for 60 seconds
Change in maximal heart rate (MaxHR) | At baseline and at 6 months
  MaxHR will be estimated using a low-risk submaximal treadmill walking test
Change in functional capacity | At baseline and at 6 months
  Functional capacity will be assessed using a movement-based screening tool titled Functional Movement Screening (FMS). The FMS will be consisted of 7 movement tasks that will be scored from 0 to 3 points and the sum will create score ranging from 0 to 21 points (0 = pain with pattern regardless of quality, 1 = unable to perform pattern, 2 = able to perform pattern with compensation/imperfection, 3 = able to perform pattern as directed).
Change in static balance | At baseline and at 6 months
  Static balance will be assessed using the Sharened Romberg test
Change in knee, hip and ankle range of motion | At baseline and at 6 months
  Knee, hip and ankle range of motion will be assessed using manual goniometer
Change in functional mobility | At baseline and at 6 months
  Functional mobility (sec) will be assessed using Gait speed test
Change in blood lipids | At baseline and at 6 months
  Total serum cholesterol (mmol/L), triglycerides (mmol/L), low density lipoprotein (mmol/L) will be measured with commercially availlable kits.
Change in muscle endurance | At baseline and at 6 months
  Muscular endurance (repetitions until muscle failure) will be assessed using timed tests (60 sec) for the abdominal musculature, upper and lower body. The tests will include partial curl-up, push-up for males and modified push-up for females (kneeling position) respectively.
Change in flexibility | At baseline and at 6 months
  Flexibility (cm) will be assessed using the modified sit-and-reach test
Change inTotal antioxidant capacity (TAC) | At baseline and at 6 months
  TAC will be will be measured with commercially available kits
Change in Cortisol | At baseline and at 6 months
  Cortisol (nmol/L) will be measured with commercially available kits
Change in insulin | At baseline and at 6 months
  Insulin (mlU/L) will be measured with commercially available kits
Change in homeostatic model assessemnet for insulin resistance (HOMA-IR) | At baseline and at 6 months
  HOMA-IR will be measured with commercially available kits. ΗΟΜΑ score will be calculated using the equation HOMA-IR = fasting insulin (mIU/L) x fasting glucose (mg/dL) / 405. HOMA-IR score will be classified using the following range: normal insulin resistance < 3, moderate insulin resistance 3-5, severe insulin resistance > 5)
Change in Interleukin 1 beta (IL-1b) | At baseline and at 6 months
  IL-1b (pg/ml) will be measured with commercially available kits
Change in Interleukin 6 (IL-6) | At baseline and at 6 months
  IL-6 (pg/ml) will be measured with commercially available kits
Change in fasting blood glucose (FBG) | At baseline and at 6 months
  FBG (mg/dL) will be measured with commercially available kits
Change in Protein Carbonyls (PC) concentration | At baseline and at 6 months
  PC (mg) will be measured in red blood cells with commercially available kits
Change in glutathione (GSH) | At baseline and at 6 months
  GSH (nmol/L) will be measured in red blood cells with commercially available kits
Change in oxidized glutathione (GSSG) | At baseline and at 6 months
  GSSG (nmol/L) will be measured in red blood cells with commercially available kits
Change in Catalase (CAT) activity | At baseline and at 6 months
  CAT activity (units) will be measured in red blood cells with commercially available kits
Change in C - reactive protein (CRP) | At baseline and at 6 months
  CRP (mg/L) will be measured with commercially available kits
Change in Uric acid (UA) | At baseline and at 6 months
  UA concentration will be measured in plasma with commercially available kits
Change in White blood cells (WBC) | At baseline and at 6 months
  White blood cells will be measured using an automatic blood analyzer
Change in Granulocyte (GRA) | At baseline and at 6 months
  GRA concentration will be measured using an automatic blood analyzer
Change in Hematocrit (HCT) | At baseline and at 6 months
  HCT concentration will be measured using an automatic blood analyzer
Change in Hemoglobin (HGB) | At baseline and at 6 months
  HGB concentration will be measured using an automatic blood analyzer
Change in red blood cells (RBC) | At baseline and at 6 months
  RBC concentration will be measured using an automatic blood analyzer
Change in Lymphocytes (LYM) | At baseline and at 6 months
  LYM concentration will be measured using an automatic blood analyzer
Change in Platelet (PLT) | At baseline and at 6 months
  PLT concentration will be measured using an automatic blood analyzer
Change in monocytes (MON) | At baseline and at 6 months
  PLT concentration will be measured using an automatic blood analyzer
Change in Cratine Kinase (CK) concentration | At 6 months and 24 hours, 48 hours and 72 hours after
  CK concentration will be measured with commercially available kits
Change in Hemoglobin A1c (HbA1c) | At baseline and at 6 months
  HbA1c concentration will be measured with commercially available kits
Change in isometric knee extensors peak torque | At baseline, at 6 months and 24 hours, 48 hours and 72 hours after
  isometric knee extensors peak torque will be assessed on an isokinetic dynamometer
Change in isometric knee flexors peak torque | At baseline, at 6 months and 24 hours, 48 hours and 72 hours after
  isometric knee flexors peak torque will be assessed on an isokinetic dynamometer
Change in eccentric knee extensors peak torque | At baseline and at 6 months
  eccentric knee extensors peak torque will be assessed on an isokinetic dynamometer
Change in eccentric knee flexors peak torque | At baseline and at 6 months
  eccentric knee flexors peak torque will be assessed on an isokinetic dynamometer
Change in concentric knee extensors peak torque | At baseline and at 6 months
  concentric knee extensors peak torque will be assessed on an isokinetic dynamometer
Change in concentric knee flexors peak torque | At baseline and at 6 months
  concentric knee flexors peak torque will be assessed on an isokinetic dynamometer
Change in counter movement jump height (CMJh) | At baseline, at 6 months and 24 hours, 48 hours and 72 hours after
  CMJh (cm) will be assessed using a force platform with each foot parallel on platform
Change in counter movement jump flight time (CMJf) | At baseline, at 6 months and 24 hours, 48 hours and 72 hours after
  CMJf (ms) will be assessed using a force platform with each foot parallel on platform
Change in counter movement jump power (CMJp) | At baseline, at 6 months and 24 hours, 48 hours and 72 hours after
  CMJp (w/kg) will be assessed using a force platform with each foot parallel on platform
Change in sprint time of 10m | At baseline, at 6 months and 24 hours, 48 hours and 72 hours after
  Sprint time (sec) will be assessed over a 10 m distance ising light cells
Change in sprint time of 30m | At baseline, at 6 months and 24 hours, 48 hours and 72 hours after
  Sprint time (sec) will be assessed over a 30 m distance ising light cells
Change in left ventricular end-diastolic volume (LVEDV) | At baseline and at 6 months
  LVEDV (ml) will be measured using echocardiography
Change in left ventricular end-systolic volume (LVESV) | At baseline and at 6 months
  LVESV (ml) will be measured using echocardiography
Change in left ventricular stroke volume (LVSV) | At baseline and at 6 months
  LVSV (ml) will be measured using echocardiography
Change in interventicular septum and systole (IVSs) | At baseline and at 6 months
  IVSs will be measured using echocardiography
Change in interventicular septum and diastole (IVSd) | At baseline and at 6 months
  IVSd will be measured using echocardiography
Change in left ventricular ejection fraction (LVEF) | At baseline and at 6 months
  LVEF (%) will be measured using echocardiography
Change in left ventricular internal diameter and diastole (LVIDd) | At baseline and at 6 months
  LVIDd (mm) will be measured using echocardiography
Change in left ventricular internal diameter and systole (LVIDs) | At baseline and at 6 months
  LVIDs (mm) will be measured using echocardiography
Change in left ventricular posterior wall end diastole (LVPWd) | At baseline and at 6 months
  LVPWd (mm) will be measured using echocardiography
Change in left ventricular mass (LV mass) | At baseline and at 6 months
  LV mass (g) will be measured using echocardiography
Change in left atrial (LA) diameter | At baseline and at 6 months
  LA diameter (mm) will be measured using echocardiography
Change in aortic root | At baseline and at 6 months
  Aortic root (mm) will be measured using echocardiography
Change in aortic valve velocity (AoV Vel) | At baseline and at 6 months
  AoV Vel (cm/s) will be measured using echocardiography
Change in aortic valve pressure gradient (AoV PG) | At baseline and at 6 months
  AoV PG (mmHg) will be measured using echocardiography
Change in right ventricular end diastole (RVD) | At baseline and at 6 months
  RVD (mm) will be measured using echocardiography
Change in right ventricular end diastole 1 (RVD1) | At baseline and at 6 months
  RVD1 (mm) will be measured using echocardiography
Change in Tricuspid Annular Plane Systolic Excursion of right ventricular functionality (TAPSE) | At baseline and at 6 months
  TAPSE (mm) will be measured using echocardiography
Change in tricuspid annular systolic velocity (TV S') of Right ventricular functionality | At baseline and at 6 months
  TV S' (mm) will be measured using echocardiography
Change in pulmonary artery systolic pressure (PASP) | At baseline and at 6 months
  PASP (mmHg) will be measured using echocardiography
Change in left ventricular fractional shortenning (FS) | At baseline and at 6 months
  Fractional shortenning (%) will be measured using echocardiography
Change in left ventricular Global Longitudinal strain (GLS) | At baseline and at 6 months
  GLS (%) will be measured using echocardiography
Change in pshycological well - being | At baseline and at 6 months
  Psychological well - being will be assessed using The General Health Questionnaire (GHQ-12) via 12 items
Change vitality | At baseline and at 6 months
  Vitality will be assessed using Subjective Vitality Scales (SVS) via 6 items. Each item is rated on a 6-point scale (1 = not at all true, 2 = not true, 3 = almost not true, 4 = almost true, 5 = true, 6 = very true). The total score ranges from 6 to 36 with a higher score indicating a better condition.
Change in motivation | At baseline and at 6 months
  E xercise behavioral will be assessed using the behavioral regulation in (BREQ-2) via 19 items questionnaire. All the 19 items were positive scored, and it was rated on a five-point for each item from 0 (not true for me) to 4 (very true for me) to identify what the participants felt about exercise.
Change in quality of life | At baseline and at 6 months
  Quality of life will be assessed using the physical and mental component subscales of the Greek 36-item Short-Form Healthy Survey (SF-36). The scores on both component subscales of the SF-36 will range from 0 to 100, with higher scores indicating better health status while the minimal clinically important difference will be 2 points.
Change in flow | At baseline and at 6 months
  Flow will be assessed using the Kurz Skala questionnaire. The Kurzskala consists 16 items which has to be answered on a seven-point rating scale from "does not apply" to "somewhat partially" to "applies".
Change in depression | At baseline and at 6 months
  Depression will be assessed using the Patient Health Questionnaire (PHQ-9), which is a self-administered instrument consisiting of 9 multiple choice questions scored from 0 to 3. Higher total scores indicate higher depression severity.

SECONDARY OUTCOMES:
Change in exercise - induced caloric expenditure | At 6 months
  Measure using portable indirect calorimetry system. Οxygen consumption will be collected during exercise session
Change in blood lactate concentration (BLa) | At 6 months
  BLa (mmol/L) concentraton will be measured in a microphotometer with commerdially available kits. Blood samples will be collected pre, mid and post execise session (single bout) at 3 minute post exercise
Change in Delay onset muscle soreness (DOMS) | At baseline, at 6 months and 24 hours, 48 hours and 72 hours after
  DOMS will be assessed using a scale consisiting of 9 multiple choices scored from 1 to 10
Change in training external load monitoring | At 6 months
  Training external load monitoring will be assessed using GPS devise
Change in training internal load monitoring | At 6 months
  Training internal load monitoring will be assessed using a pulse devises
Body Height | At baseline
  Height (cm) will be measured using stadiometer
Electrocardiogram (ECG) | At baseline
  ECG will be recorded using the electrical heart signals by electrocardiogram device in order to examined the resting heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis G Fatouros, Prof, Study Director — University of Thessaly
Locations (1):
- University o Thessaly, School of Physical Education and Sports Science, Trikala, Greece